CLINICAL TRIAL: NCT06497608
Title: Exploring the Cellular and Molecular Mechanisms of the Development and Progression of Diabetic Retinopathy Based on Single-cell Sequencing
Brief Title: Single-Cell Insights Into Diabetic Retinopathy Mechanisms
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi Zheng, Prof., Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 2023321
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — We will collect retinal samples from 3 patients with advanced proliferative diabetic retinopathy who underwent prosthetic eye implantation, as well as retinal samples from 3 healthy cadaver donors. Additionally, we will collect aqueous humor, vitreous fluid, and plasma samples from 30 patients undergoing diabetic retinopathy surgery and 30 macular hole surgery patients without diabetic retinopathy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- scRNA_DR: Patients with proliferative diabetic retinopathy who underwent prosthetic eye implantation.
- scRNA_normal: Body donors without history of diabetic retinopathy
- Validate_DR: Patients with proliferative diabetic retinopathy (PDR) who underwent vitrectomy surgery
- Validate_normal: Patients who underwent vitrectomy surgery for macular hole (MH) and did not have diabetic retinopathy (DR)

SUMMARY:
This study aims to uncover the cellular and molecular mechanisms of diabetic retinopathy through single-cell sequencing to identify new therapeutic targets.

The study will collect retinal tissue samples from 3 patients with advanced proliferative diabetic retinopathy who underwent prosthetic eye implantation and 3 normal cadaver donors. Additionally, aqueous humor, vitreous fluid, and plasma samples from patients with severe diabetic retinopathy requiring surgery and macular hole surgery patients without diabetic retinopathy will be analyzed using ELISA, qPCR, and Western Blot. These experiments will validate sequencing results and explore the pathogenesis of diabetic retinopathy to identify potential treatment targets.

DETAILED DESCRIPTION:
Diabetic retinopathy is the leading cause of blindness among the working population worldwide. However, its pathogenesis is not fully understood, and effective prevention and treatment methods are limited. This study, initiated by Shanghai First People's Hospital, aims to explore the cellular and molecular mechanisms underlying its occurrence through methods such as single-cell sequencing, to identify new intervention targets. This study plans to collect retinal tissue samples from 3 patients each who underwent prosthetic eye implantation due to late-stage proliferative diabetic retinopathy blindness and from 3 normal cadaver donors at the Ophthalmology Department of Shanghai First People's Hospital for single-cell sequencing and bioinformatics analysis. Additionally, samples of aqueous humor, vitreous fluid, and plasma will be collected from 30 patients with severe diabetic retinopathy requiring surgery and from 30 macular hole surgery patients without diabetic retinopathy. These samples will be subjected to experiments such as ELISA, qPCR, and Western Blot to validate sequencing results, investigate the pathogenesis of diabetic retinopathy, and identify potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria :

* For the single-cell sequencing group: Patients with advanced proliferative diabetic retinopathy (PDR) resulting in blindness or ocular atrophy, who voluntarily opt for enucleation and ocular prosthesis implantation surgery, and have no systemic or local contraindications to surgery. For the validation group: patients with severe PDR lesions requiring vitrectomy, and who also have no systemic or local contraindications to surgery.
* Patients who voluntarily agree to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

* Patients with severe systemic diseases such as autoimmune diseases or cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit the Department of Ophthalmology at Shanghai General Hospital and meet the inclusion and exclusion criteria of this study.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Single cell sequencing result | 1 month
  Single cell RNA and ATAC sequencing of human retinas

SECONDARY OUTCOMES:
Validation experiment result | 1 month
  Experiments such as ELISA and immunofluorescence staining to validate the result from single cell sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Zheng, Prof., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided
Due to the confidentiality policy of the Chinese National Health Council and institutional patient privacy regulations, we have not decided on the plan to share IPD. However, the data are available from the corresponding authors upon request.

REFERENCES:
- [Background] Hu Z, Mao X, Chen M, Wu X, Zhu T, Liu Y, Zhang Z, Fan W, Xie P, Yuan S, Liu Q. Single-Cell Transcriptomics Reveals Novel Role of Microglia in Fibrovascular Membrane of Proliferative Diabetic Retinopathy. Diabetes. 2022 Apr 1;71(4):762-773. doi: 10.2337/db21-0551. PMID 35061025
- [Background] Niu T, Fang J, Shi X, Zhao M, Xing X, Wang Y, Zhu S, Liu K. Pathogenesis Study Based on High-Throughput Single-Cell Sequencing Analysis Reveals Novel Transcriptional Landscape and Heterogeneity of Retinal Cells in Type 2 Diabetic Mice. Diabetes. 2021 May;70(5):1185-1197. doi: 10.2337/db20-0839. Epub 2021 Mar 5. PMID 33674409
- [Background] Van Hove I, De Groef L, Boeckx B, Modave E, Hu TT, Beets K, Etienne I, Van Bergen T, Lambrechts D, Moons L, Feyen JHM, Porcu M. Single-cell transcriptome analysis of the Akimba mouse retina reveals cell-type-specific insights into the pathobiology of diabetic retinopathy. Diabetologia. 2020 Oct;63(10):2235-2248. doi: 10.1007/s00125-020-05218-0. Epub 2020 Jul 30. PMID 32734440
- [Background] Ziegenhain C, Vieth B, Parekh S, Reinius B, Guillaumet-Adkins A, Smets M, Leonhardt H, Heyn H, Hellmann I, Enard W. Comparative Analysis of Single-Cell RNA Sequencing Methods. Mol Cell. 2017 Feb 16;65(4):631-643.e4. doi: 10.1016/j.molcel.2017.01.023. PMID 28212749
- [Background] Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010 Jul 10;376(9735):124-36. doi: 10.1016/S0140-6736(09)62124-3. Epub 2010 Jun 26. PMID 20580421